CLINICAL TRIAL: NCT01652963
Title: Evaluating a Picture-based Computerised Assessment and Training Paradigm for Cognitive Behaviour Therapy Skills in Adults With Intellectual Disabilities
Brief Title: Picture-based Computerised Assessment and Training of Cognitive Behaviour Therapy Skills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: UEA-6345832-MED1; 12/EE/0284 (Other: NHS REC Hertfordshire)
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Intellectual Disabilities
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control task (No Intervention): The no-intervention control task consists of a presentation of the stimuli used in the training task. Participants will see situations and listen to the simultaneous voice recordings. Unlike in the training task participants will not receive instructions to link situations and emotions. There is no task requirement, just a presentation of the situation stimuli to assure that potential training effects are due to the training programme and not merely to the presentation of scenarios. The duration of the presentation of stimulus materials in the control group will range between fifteen and thirty minutes. The variable duration is necessary so the primary investigator cannot assume a participant's intervention group based on the duration of the intervention task.
- Reed and Clements Training Task (Experimental): The training task consists of 2 blocks of 6 items with items presented randomly within each block and blocks being counterbalanced between participants. Block 1 presents a situation and prompts participants to identify whether they would feel happy or sad in the given situation. Block 2 presents an emotion (happy or sad) and prompts the participant to identify which of two situations (positive or negative) most likely preceded this emotion. Within each block there will be at least one and maximum three training rounds. The second and third training rounds will only consist of the items to which the participant responded incorrect in the previous round. Each item in rounds 2 and 3 will be followed by feedback.
  Interventions: Other: Reed and Clements Training Task

INTERVENTIONS:
Other: Reed and Clements Training Task — see study arm: Reed and Clements Training Task. Training task developed to improve cognitive mediation skills in people with intellectual disabilities.
  Arms: Reed and Clements Training Task

SUMMARY:
The proposed research aims to investigate whether people with intellectual disabilities are able to understand and apply the theoretical principles of cognitive behaviour therapy (CBT) regarding the interaction between events, beliefs and emotions. Two studies are designed to assess and train the ability to link events, beliefs and emotions.

Study 1 pilots computer-based tasks to assess the ability to link events, beliefs and emotions as well as a computer-based training programme aimed to link events and emotions. Task and training stimuli will be presented by line drawings to investigate whether a picture-based approach can reduce the impact of verbal ability on task performance. Training effectiveness is evaluated compared to a no-training control task.

Study 2 compares the line drawings-based approach of Study 1 to a photographic approach to investigate whether the use of photographs can increase training effectiveness and further reduce the impact of verbal ability. It is hypothesised that the high reality value of photographic task stimuli, as compared to line drawings, will have positive effects on the assessment and training of CBT skills. It is anticipated that the findings of this research will improve our ability to help people with intellectual disabilities receive CBT.

DETAILED DESCRIPTION:
STUDY 1

HYPOTHESES

1. A picture-based training programme aimed to link situations and emotions improves the cognitive behaviour therapy (CBT) skill of linking situations, beliefs and emotions.
2. People with intellectual disabilities can understand and follow the procedures for computer based assessment and training tasks.

DESIGN A 2 x (2 x S) mixed experimental design will be used with a between-subjects factor (Intervention: training group versus control group) and a within-subjects factor (Time: baseline assessment versus post-intervention assessment). Baseline and post-intervention assessment of CBT skills will be derived from the cognitive mediation task developed by Dagnan et al. (2000). Performance on the post-intervention assessment is considered the primary outcome variable of the study (Hypothesis 1).

The intervention in the training group will be based on the Reed and Clements task (1989) which assesses the ability to link situations and emotions. The intervention in the control group will consist of the presentation of the same stimulus materials as the intervention group. The materials will be presented without specific training instructions and matched in time with the duration of the training group intervention. The control group intervention allows for an evaluation of training task efficacy rather than evaluating the confounding effects of presenting certain stimulus materials.

Assessment and training tasks will all be conducted individually and they will be presented via a computer programme on a laptop computer with an external response box (Hypothesis 2).

PROCEDURES

Pre-study procedures. When consent has been obtained, the principal investigator assesses verbal ability (BPVS-2) and level of intellectual functioning (WASI-II). Participants who meet the inclusion criteria will then be invited to complete the baseline assessments.

Baseline assessments. At baseline, the researcher will introduce the laptop computer and the external response box. The computer program will be introduced and one sample item of the assessment will be solved by the computer to illustrate how the task works. The sample item will then be repeated for the participant to solve and for the researcher to check if the participant understands the procedures of the task. The sample item will be repeated until the participant understands the procedures and will have learned how to operate the response box. The primary investigator will be present to assist the participant with the use of the response box and to explain the task procedures.

The adapted cognitive mediation task consists of two blocks of twelve exercises. Exercises are randomised within each block and blocks are counterbalanced between participants. Block 1 presents the six scenarios paired once with a positive and once with a negative thought resulting in twelve task items. Each task item presents two pictures of a situation followed by a picture of a positive or negative thought about this situation. Participants are then prompted to identify which of two pictured emotions (happy or sad) they would feel following the given situation and thought. Block 2 presents each scenario paired with a positive and negative emotional response to create twelve task items. Each item presents two pictures of a situation followed by a picture of an emotional response (happy or sad). Participants are then prompted to identify which of two thoughts (positive or negative) is most likely to cause the given emotion in the presented situation.

Intervention in training group. Participants will be given a break between the baseline assessment and the intervention task. The primary investigator will be replaced by a second researcher who will be responsible for conducting the intervention task. The intervention in the training group is based on a task developed by Reed and Clements (1989). The training task consists of two blocks of six items presented randomly within each block and blocks being counterbalanced between participants. Block 1 follows the original task by presenting a situation and prompting participants to identify whether they would feel happy or sad in the given situation. Block 2 presents an emotion (happy or sad) and prompts the participant to identify which of two situations (positive or negative) most likely preceded this emotion. Each block contains three positive (positive situation or happy emotion given) and three negative items (negative situation or sad emotion given). The training task will begin with a sample exercise solved by the computer and a sample exercise for the participant, similarly to the procedures for the baseline assessment. Within each block there will be at least one and maximum three training rounds. In the first training round all six items within a block will be presented. The second and third training rounds will only consist of the items to which the participant responded incorrect in the previous round. Each item will now be followed by feedback and incorrect responses will be followed by the correct response.

Intervention in control group. The intervention in the control group consists of a presentation of the stimuli used in the training task. Participants will see situations and listen to the simultaneous voice recordings. Unlike in the training task participants will not receive instructions to link situations and emotions. There is no task requirement, just a presentation of the situation stimuli to assure that potential training effects are due to the training programme and not merely to the presentation of scenarios. The duration of the presentation of stimulus materials in the control group will range between fifteen and thirty minutes. The variable duration is necessary so the primary investigator cannot assume a participant's intervention group based on the duration of the intervention task.

Post-intervention assessment. Post-intervention assessments will take place fifteen minutes after the intervention task. The second researcher leaves the room as the primary investigator returns to conduct the post-intervention assessments. Participants will be reminded to not disclose any information concerning the intervention task with the researcher. The post-intervention assessment consists of the adapted cognitive mediation task of the baseline assessment. The same procedures of the baseline assessment apply to the post-intervention assessment. Within each block of six exercises, four exercises will be randomly chosen from the baseline items and two new items will be added.

STUDY 2

HYPOTHESES

1. Photographs may have an advantage over standard line drawings to improve performance on tasks assessing the ability to link situations, beliefs and emotions. It is hypothesised that a photographic approach will increase effectiveness of the CBT skills training. It is assumed that the high reality value of photographs may enhance identification with the task materials and thereby improve performance.
2. A photographic approach may, when compared to the standard verbal approach and a line drawings-based approach, reduce the impact of verbal ability on the assessment of CBT skills.
3. A CBT training programme aimed to link situations and emotions may improve both emotion recognition skills and cognitive mediation skills (as assessed by the ability to link situation, beliefs and emotions).

DESIGN

Study 2 is based on a 2 x (2 x S) mixed experimental design with a between-subjects factors (Training group: line drawings group versus photographs group) and a within-subjects factor (Time: baseline assessment versus post-intervention assessments).

Baseline and post-intervention assessment of CBT skills will consist of the adapted cognitive mediation task, as it is used and described in Study 1, and of an emotion recognition task. Both assessments will have line drawings and photographs as stimulus materials to investigate Hypotheses 1 and 3.

The intervention in both training groups will be based on the Reed and Clements task (1989) as described in Study 1. Participants in the line drawings group will receive the adapted Reed and Clements task (1989) based on line drawings. Participants in the photographs group will be presented photographs as task stimuli. The content of the task items does not differ between the training groups, only the pictorial presentation of the items differs (Hypothesis 1 and 2). There will be no separate control group.

PROCEDURES

Pre-study procedures. These procedures are identical to the pre-study procedures described in Study 1.

Baseline assessments. The primary investigator will begin by reminding the participant that their participation is voluntary, that all data will be anonymous and that they have the right to withdraw from the study at any time. The researcher will then introduce the laptop computer and the external response box and will continue to explain the procedures for the task.

Baseline assessment will consist of the counterbalanced presentation of the emotion recognition task and the adapted cognitive mediation task. The computer program will be introduced and one sample item of the first assessment will be solved by the computer to illustrate how the task works. The sample item will then be repeated for the participant to solve and for the researcher to check if the participant understands the procedures of the task. The sample item will be repeated until the participants understands the procedures and will have learned how to operate the response box. Baseline assessment will consist of the counterbalanced presentation of the emotion recognition task and the adapted cognitive mediation task. For each task half of the items will be presented in line drawings and half of the items in photographs. The procedures for the adapted cognitive mediation task have been described in Study 1.

The emotion recognition task in Study 2 will consist of two blocks of six exercises, counterbalanced between participants. The exercises of block 1 are based on line drawings and the exercises of block 2 are based on photographs. All exercises, regardless of the block condition, will begin with a three second presentation of a happy face or a sad face. A voice recording will be played telling participants which emotion is pictured. This presentation will be followed by a one second blank screen. Following the blank screen, three new pictures of various emotions will be shown. A recorded voice will prompt the participants to identify which of the three presented emotions is similar to the initially presented emotion. The target emotions will be happy and sad, while the two distracter emotions may vary between neutral, annoyed, disgusted, grumpy, surprised and angry.

Intervention. Participants will be given a break between the baseline assessments and the training task. The primary investigator will leave the room and will be replaced by the second researcher who will be responsible for conducting the training task. The training task is the adapted Reed and Clements (1989) task based on line drawings for the line drawings group and on photographs for the photographs group. The procedures follow the procedure of this training task in Study 1.

Post-intervention assessments. After the training task participants will be given a short break and the principal investigator will return to conduct the post-intervention assessments. The researcher will remind participants to not disclose any information regarding the training task. Post-intervention assessment of the adapted cognitive mediation task and the emotion recognition task will follow the same procedures as for their baseline assessment. For the post-intervention assessment half of the baseline items within each task block will be replaced with new items to control for rehearsal effects and test for generalisation of training effects to new items.

ELIGIBILITY:
Inclusion Criteria:

* Intellectual disability

Exclusion Criteria:

* Visual impairments
* Auditory impairments
* Currently receiving cognitive behaviour therapy
* Acute psychosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Cognitive mediation skills | 15 minutes at baseline
  The primary outcome measure is the ability to link situations, beliefs and emotions assessed by the adapted ABC task. This task is based on the cognitive mediation task developed by Dagnan, Chadwick and Proudlove (2000). Performance on the post-intervention assessment will be compared to baseline assessment for the control group and the training group in Study 1, and for the line drawings-based and the photograph-based training group in Study 2.

SECONDARY OUTCOMES:
Emotion recognition skills | 15 minutes at baseline
  Computer-based task assessing emotion recognition skills.

OTHER OUTCOMES:
feasibility of computer-based tasks | 1 hr, baseline, intervention, post-assessment
  Feasibility of computer-based tasks will be measured by the type and number of assisting interventions by the researchers and the frequency of repeating the sample items of each task.

CONTACTS AND LOCATIONS:
Overall Officials: Leen Vereenooghe, BSc, MSc, Principal Investigator — University of East Anglia
Locations (3):
- United Kingdom (3):
  - NCH&C NHS Trust Learning Disability Services, Norwich, Norfolk
  - Nansa, Norwich, Norfolk
  - Genesis - Orwell Mencap, Ipswich, Suffolk